CLINICAL TRIAL: NCT06029725
Title: RFMN in Combination With 1927 nm Thulium Laser for Treating Photoaged Skin: a Prospective, Controlled Study
Brief Title: RFMN in Combination With 1927 nm Thulium Laser for Treating Photoaged Skin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Lynhda Nguyen, Principle Investigator, Universitätsklinikum Hamburg-Eppendorf
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-23
Record Dates: First submitted 2023-08-23; First posted 2023-09-08 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Photoaging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RFMN+Thulium (Active Comparator)
  Interventions: Device: radiofrequency microneedling combined with 1927 nm thulium laser
- RFMN (Active Comparator)
  Interventions: Device: radiofrequency microneedling monotherapy

INTERVENTIONS:
Device: radiofrequency microneedling combined with 1927 nm thulium laser — 1. session: radiofrequency microneedling + 1927 nm thulium laser
  2. session: 1927 nm thulium laser monotherapy
  3. session: 1927 nm thulium laser monotherapy
  Arms: RFMN+Thulium
Device: radiofrequency microneedling monotherapy — 1 session: radiofrequency microneedling monotherapy
  Arms: RFMN

SUMMARY:
The appearance of the aging skin is influenced by different factors including by the reduced elasticity and increased laxity of the skin, the decreasing volume as well as pigmentation disorders and dilated vascular markings. Currently, there are different methods available to treat the aging skin. Here, the combined treatment of radiofrequency micro needling (RFMN) and thulium laser has been commonly used in clinical practice.

The aim of this clinical study is to investigate the efficacy, patient satisfaction, safety of RFMN and thulium laser treatment in patients with facial, age-related skin laxity, wrinkles, and pigmented lesions.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from the age of 30 years
* good general condition, no relevant previous diseases
* Presence of wrinkles, dermatochalasis on the face, pigment spots, which are an indication for RFMN and thulium laser or comparable methods
* Cognitive ability and willingness to give consent (informed consent)
* Be willing and able to attend follow-up visits

Exclusion Criteria:

* Age < 30 years
* Pregnancy or breastfeeding
* Excessive subcutaneous fatty tissue under the cheeks
* Significant scarring of the region to be treated
* open wounds or lesions of the region to be treated
* Severe or cystic facial acne
* Metallic implants in the face or neck region
* Mental illnesses (psychoses, body perception disorders)
* Use of isotretinoin or other retinoids, psychotropic drugs, coumarins or heparins in the last 2 weeks
* Fillers in the region to be treated < 4 weeks prior and during the study period
* Resurfacing (fractional, ablative, nonablative) of the region of interest < 2 months prior and during the study period
* Plastic aesthetic procedures or other surgical procedures < 6 months prior and during the study period
* Tendency to have excessive scarring
* Lack of informed consent

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in wrinkles | 6 months after last treatment session
  software-assisted evaluation of wrinkles (Vectra(R) Software, Canfield)
Change in volume | 6 months after last treatment session
  software-assisted evaluation of volume (Vectra(R) Software, Canfield)
Change in pigmentation | 6 months after last treatment session
  software-assisted evaluation of pigmentation (Vectra(R) Software, Canfield)

SECONDARY OUTCOMES:
Pain intensity | 10 minutes after starting each treatment session, one treatment session takes 30-50 minutes
  pain intensity (numeric rating scale) during treatment
Adverse Events | before every treatment session, at every follow-up visit (3 and 6 months post-treatment)
  number of adverse events (AE)
Withdrawals due to AE | before every treatment session, at every follow-up visit (3 and 6 months post-treatment)
  number of withdrawal due to AE

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berneburg M, Plettenberg H, Krutmann J. Photoaging of human skin. Photodermatol Photoimmunol Photomed. 2000 Dec;16(6):239-44. doi: 10.1034/j.1600-0781.2000.160601.x. PMID 11132125
- [Background] el-Domyati M, el-Ammawi TS, Medhat W, Moawad O, Brennan D, Mahoney MG, Uitto J. Radiofrequency facial rejuvenation: evidence-based effect. J Am Acad Dermatol. 2011 Mar;64(3):524-35. doi: 10.1016/j.jaad.2010.06.045. PMID 21315951
- [Background] Zelickson BD, Kist D, Bernstein E, Brown DB, Ksenzenko S, Burns J, Kilmer S, Mehregan D, Pope K. Histological and ultrastructural evaluation of the effects of a radiofrequency-based nonablative dermal remodeling device: a pilot study. Arch Dermatol. 2004 Feb;140(2):204-9. doi: 10.1001/archderm.140.2.204. PMID 14967794
- [Background] Nguyen L, Blessmann M, Schneider SW, Herberger K. Radiofrequency Microneedling for Skin Tightening of the Lower Face, Jawline, and Neck Region. Dermatol Surg. 2022 Dec 1;48(12):1299-1305. doi: 10.1097/DSS.0000000000003607. Epub 2022 Sep 29. PMID 36449871
- [Background] Wang JV, Christman MP, Feng H, Ferzli G, Jeon H, Geronemus RG. Laser-assisted delivery of tranexamic acid for melasma: Pilot study using a novel 1927 nm fractional thulium fiber laser. J Cosmet Dermatol. 2021 Jan;20(1):105-109. doi: 10.1111/jocd.13817. Epub 2020 Nov 11. PMID 33174686
- [Background] Lu K, Cai S. Efficacy and safety comparison between 1927 nm thulium laser and 2940 nm Er:YAG laser in the treatment of facial atrophic acne scarring: a prospective, simultaneous spilt-face clinical trial. Lasers Med Sci. 2022 Apr;37(3):2025-2031. doi: 10.1007/s10103-021-03465-0. Epub 2021 Nov 26. PMID 34826022
- [Background] Serra M, Bohnert K, Sadick N. A randomized, single-blind, study evaluating a 755-nm picosecond pulsed Alexandrite laser vs. a non-ablative 1927-nm fractionated thulium laser for the treatment of facial photopigmentation and aging. J Cosmet Laser Ther. 2018 Oct;20(6):335-340. doi: 10.1080/14764172.2018.1493513. Epub 2018 Jul 18. PMID 30019970
- [Background] Friedman PM, Dover JS, Chapas A, Rahman Z, Ross EV, Kilmer SL, Roberts WE, Sodha P, Stimmel JB, Moncrief MBC, Waibel JS. 1,550 nm Erbium-Doped and 1,927 nm Thulium Nonablative Fractional Laser System: Best Practices and Treatment Setting Recommendations. Dermatol Surg. 2022 Feb 1;48(2):195-200. doi: 10.1097/DSS.0000000000003321. PMID 35050945
- [Derived] Nguyen L, Blessmann M, Schneider SW, Herberger K. Radiofrequency Microneedling With 1927 nm Thulium Laser Versus Radiofrequency Microneedling Monotherapy for Rejuvenation of Photoaged Skin. J Cosmet Dermatol. 2026 Jan;25(1):e70685. doi: 10.1111/jocd.70685. PMID 41566557